CLINICAL TRIAL: NCT04439409
Title: AVASNA : Variability of the Autonomic Nervous System (ANS) During Cluster Headache (CH).
Brief Title: Variability of the Autonomic Nervous System (ANS) During Cluster Headache (CH).
Acronym: AVASNA
Status: Terminated | Type: Observational
Why Stopped: No inclusions for 2 years
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 19CH103; 2019-A01343-54 (Other: ANSM)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-04

CONDITIONS: Cluster Headache
Keywords: Cluster Headache; Autonomic Nervous System; Seizure; Holter; Electrocardiogram; (LF/HF) ratio; Daytime seizure; Night seizure
MeSH Terms: conditions — Cluster Headache; Seizures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Cluster Headache (CH): Patients with Cluster Headache (CH) will be included. They will have a Holter electrocardiogram during 7 days.
  Interventions: Device: Holter electrocardiogram

INTERVENTIONS:
Device: Holter electrocardiogram — Holter electrocardiogram will be carried during 7 days to measure heart's electrical activity continuously.

SUMMARY:
Cluster Headache (CH) is associated with ipsilateral vegetative signs, related to parasympathetic system hyperactivity and/or signs of sympathetic hypoactivity. The precise mechanism of Cluster Headache (CH) is still unknown. The question is whether these dysautonomic disorders are simply secondary to the Cluster Headache (CH) process or whether they are the triggering factor.

DETAILED DESCRIPTION:
This study cares about the evolution of the Autonomic Nervous System (ANS) in Cluster Headache (CH) seizures. Patients will be offered Holter ECG to study the temporal relationships between changes in Autonomic Nervous System (ANS) activity during Headache (CH) seizures and changes in Autonomic Nervous System (ANS) activity before and after seizure treatment, using heart rate variability measurement.

The hypothesis is that there would be an initial temporary sympathetic activation, followed quickly by parasympathetic hyperactivation and a return to a state of equilibrium.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Affiliated or entitled to a Social Security scheme
* Resident in the territories of the hospital grouping of Loire territory (located less than 50 km away)
* Whose diagnosis of episodic or chronic Cluster Headache (CH) has been confirmed according to International Classification of Headache Disorders (ICHD)- 3 criteria
* With a regular sinus rhythm and heart rate

Exclusion Criteria:

* Conditions contraindicating the use of injectable sumatriptan
* Conditions likely to affect the Autonomic Nervous System (ANS): dysautonomic sensory neuropathies, sleep apnea syndrome, etc.
* Cognitive or language disorders that may interfere with pain assessment and seizure follow-up.
* Patients taking treatments that may modify the Autonomic Nervous System (ANS): catecholamine (adrenaline, noradrenaline, dopamine), B-stimulants (isoprenaline, dobutamine, dopexamine, salbutamol, terbutaline, fenoterol, orciprenaline, clenbuterol, salmeterol, formoterol), B-blockers, alpha-stimulants (midodrine, alpha-methyl-dopa, clonidine, rilmenidine, moxonidine), alpha-blockers (phentolamine, prazosin, urapidil), amphetamine, tyramine, ephedrine, selegiline, cocaine, imipramine.
* Impossibility to submit to the medical follow-up of the program for geographical, social or psychological reasons.
* Patient deprived of liberty or under guardianship.
* Patient with preventive background treatment of Cluster Headache (CH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cluster Headache (CH) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Low Frequency/High Frequency (LF/HF) ratio at the onset of the first night seizure | Day: 7
  Comparison of the Low Frequency/High Frequency (LF/HF) ratio at the onset of the first night seizure during the basal period, pre-seizure, seizure and after the seizure.

SECONDARY OUTCOMES:
Low Frequency/High Frequency (LF/HF) ratio at the onset of the first daytime seizure | Day: 7
  Comparison of the Low Frequency/High Frequency (LF/HF) ratio at the onset of the first daytime seizure during the basal period, pre-seizure, seizure and after the seizure.
Low Frequency during daytime and night seizure | Day: 7
  Comparison of measure of Low Frequency during daytime and night seizure.
High Frequency (HF) during daytime and night seizure | Day: 7
  Comparison of measure of High Frequency (HF) during daytime and night seizure.
Correlation between several parameters | Day: 7
  Correlation between Heart Rate Variability (HRV), changes in the Low Frequency/High Frequency (LF/HF) ratio, the Low Frequency (LF) and the High Frequency (HF), and the intensity of pain measured on the Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Christelle CREAC'H, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No